CLINICAL TRIAL: NCT00670462
Title: Maintenance-Tailored Obesity Treatment
Acronym: LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0402S56276; R01DK067362 (NIH)
Record Dates: First submitted 2008-04-30; First posted 2008-05-01 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Obesity
Keywords: obesity, weight loss, treatment
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Behavioral Treatment (SBT) (Active Comparator): Standard Behavioral Treatment (SBT) for weight loss intervention introduces a core set of instructions on diet and exercise at the beginning of the intervention and then "embellishes" these instructions with suggested refinements of behavioral choices over time (e.g., different menus and amounts or types of physical activity).
  Interventions: Behavioral: Standard Behavioral Treatment (SBT)
- Maintenance-Tailored Treatment (MTT) (Experimental): Maintenance-Tailored Treatment (MTT) for weight loss intervention treats diet and exercise strategy "embellishments" as separate interventions with discrete and independent status. MTT differs from SBT in its emphasis on skills for long-term weight control, namely, the strategy of initiating varied weight-control strategies as a response to the demands of changing environmental challenges and to sustain effective cues and reinforcements needed to motivate weight-loss behaviors.
  Interventions: Behavioral: Maintenance-Tailored Treatment (MTT)

INTERVENTIONS:
Behavioral: Standard Behavioral Treatment (SBT) — SBT is state-of-the-art behavioral weight loss treatment, comprised of 6 months of weekly treatment meetings followed by 6 months of biweekly meetings and 6 months of monthly meetings. Topical coverage and behavioral assignments include typical combination of energy balance information and self-control skills training. MTT has the same number of treatment contacts, but the contacts are distributed in distinct 8-week segments, each of which have a unique topic and unique behavioral assignments. Between each segment, participants are left on their own for 4 weeks with instructions to continue regular weighing but otherwise to make their own choices about what to do for weight control.
  Other Names: lifestyle intervention
  Arms: Standard Behavioral Treatment (SBT)
Behavioral: Maintenance-Tailored Treatment (MTT)
  Arms: Maintenance-Tailored Treatment (MTT)

SUMMARY:
This study is a randomized clinical trial comparing state-of-the-art, standard behavior therapy for weight loss (SBT) with a maintenance tailored treatment (MTT) with varied behavioral prescriptions, goals, and formats over time. The overall hypothesis in the study is that the two treatment approaches will show different patterns of weight loss over time, and in particular that the MTT approach would be associated with better long-term maintenance of weight loss.

DETAILED DESCRIPTION:
Recent dramatic increases in prevalence have made obesity the number one nutritional problem in the US. Of particular concern is the fact that, although available treatments are effective in producing clinically significant weight loss, their ability to sustain weight loss long term is poor. This study is based on a conceptual analysis of this problem that argues for greater attention to two issues related to the temporal dynamics of the challenge of long-term weight control. These are: 1) the environment is continually changing and is not supportive of weight control and 2) the intervention methods that are effective in inducing short-term changes in behaviors and weight often lose their potency over time because of habituation.

This study is a randomized trial in which obese men and women are assigned to one of two study conditions, Standard Behavior Treatment (SBT) or Maintenance-Tailored Treatment (MTT). The MTT has adaptation to change as its central theme. A primary technique that is used to convey this theme that is different than traditional behavior treatment is that participants are asked to deliberately change weight-loss strategies systematically over time rather than to use the same approach consistently across time. Frequent change serves as a platform for teaching a larger variety of weight-control skills and thus strengthening study participants ability to adapt their weight-control strategies to changing circumstances. Changing weight-control strategies regularly also helps to reduce the extent to which habituation to strategies implemented invariantly over time diminish the salience of behavioral cues and the potency of behavioral reinforcers for sustaining weight-control efforts over time. Individuals in both treatment groups receive active intervention for a period of 18 months, followed by 12 months of no-treatment follow-up.

The primary hypothesis tested is that MTT will produce larger mean weight losses at 30-month follow-up than SBT. Moreover, it is predicted that the better long-term success of the MTT group will be due primarily to better weight-loss success beyond 6 months, the point at which most people begin to regain weight with standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Body mass index between 30.0 and 37.0

Exclusion Criteria:

* serious current physical disease (e.g., heart disease, cancer, and diabetes) for which physician supervision of diet and exercise would be needed.
* initial fasting glucose values above 120 mg/dl
* resting blood pressure at or above 90 DBP or 150 SBP will be strongly encouraged to see their primary care physician for further evaluation and will not be accepted into the study unless they do so and have physician consent for participation.
* physical problems that preclude their participation in the diet and exercise components of the program
* currently taking weight-loss medications
* currently participating in another formal weight loss-program
* currently pregnant or plan to become pregnant during the next 30 months
* currently receiving treatment for a major psychological disorder or have scores on the Beck Depression Inventory above 27.0, indicative of likely clinical depression.
* only one individual per household accepted into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2004-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Jeffery, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, School of Public Health, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Behavioral Treatment (SBT): Standard Behavioral Treatment (SBT) for weight loss introduces a core set of instructions on diet and exercise at the beginning of the intervention and then "embellishes" these instructions with suggested refinements of behavioral choices over time (e.g., different menus and amounts or types of physical activity).
  weight loss intervention: SBT is state-of-the-art behavioral weight loss treatment, comprised of 6 months of weekly treatment meetings followed by 6 months of biweekly meetings and 6 months of monthly meetings. Topical coverage and behavioral assignments include typical combination of energy balance information and self-control skills training.
- Maintenance-Tailored Treatment (MTT): Maintenance-Tailored Treatment (MTT) for weight loss treats diet and exercise strategy "embellishments" as separate interventions with discrete and independent status. MTT differs from SBT in its emphasis on skills for long-term weight control, namely, the strategy of initiating varied weight-control strategies as a response to the demands of changing environmental challenges and to sustain effective cues and reinforcements needed to motivate weight-loss behaviors.
  weight loss intervention: MTT has the same number of treatment contacts, but the contacts are distributed in distinct 8-week segments, each of which have a unique topic and unique behavioral assignments. B
Period: Overall Study
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Started | 106 | 107
Completed | 76 | 76
Not Completed | 30 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT) | Total
Number analyzed (Participants) | 106 | 107 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (10.6) | 48.5 (10.5) | 48.8 (10.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 103 | 205
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 51 | 49 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 29 | 50
  White | 74 | 69 | 143
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 106 | 107 | 213
energy intake (kcal/day) [Mean (Standard Deviation); unit: kcal/day] | 1980.4 (924.7) | 1976.4 (922.7) | 1978.4 (921.5)
energy expenditure (kcal/wk) [Mean (Standard Deviation); unit: kcal/wk] | 884.2 (958.7) | 954.2 (1267.2) | 919.2 (1112.95)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 35.2 (2.8) | 34.6 (2.8) | 34.9 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Time Frame: Baseline to18 months
Population: Waist-to-hip Ratio" was assessed for all Males and Females, separately, irrespective of the intervention to which participants were randomized.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 106 | 107
kg | 9.3 (8.8) | 8.3 (8.9)

2. Secondary Outcome: Physical Activity, Energy Expenditure
Description: change from baseline in energy expenditure at 6 months
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kcal/wk
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 98 | 101
kcal/wk | 964.1 (131.8) | 726.4 (128.2)

3. Secondary Outcome: Change From Baseline in Energy Intake at 6 Months
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 98 | 101
kcal/day | -491.2 (72.6) | -576.4 (71.1)

4. Secondary Outcome: Blood Pressure
Time Frame: baseline, 6, 12, 18, and 30 months
Reporting Status: Not Posted

5. Secondary Outcome: Waist-to-hip Ratio at Baseline
Time Frame: baseline
Measure: Mean (Standard Error); unit: ratio
Groups:
- Women SBT and MTT; Men SBT and MTT: Standard Behavioral Treatment (SBT) for weight loss introduces a core set of instructions on diet and exercise at the beginning of the intervention and then "embellishes" these instructions with suggested refinements of behavioral choices over time (e.g., different menus and amounts or types of physical activity).
  Maintenance-Tailored Treatment (MTT) for weight loss treats diet and exercise strategy "embellishments" as separate interventions with discrete and independent status. MTT differs from SBT in its emphasis on skills for long-term weight control, namely, the strategy of initiating varied weight-control strategies as a response to the demands of changing environmental challenges and to sustain effective cues and reinforcements needed to motivate weight-loss behaviors.
Arm/Group | Women SBT and MTT | Men SBT and MTT
Number analyzed (Participants) | 113 | 100
ratio | .85 (.01) | .99 (.01)

6. Secondary Outcome: Blood Glucose
Time Frame: baseline, 6, 12, 18, and 30 months
Reporting Status: Not Posted

7. Secondary Outcome: Insulin
Time Frame: baseline, 6, 12, 18, and 30 months
Reporting Status: Not Posted

8. Secondary Outcome: HDL
Time Frame: baseline, 6, 12, 18, and 30 months
Reporting Status: Not Posted

9. Secondary Outcome: Triglycerides
Time Frame: baseline, 6, 12, 18, and 30 months
Reporting Status: Not Posted

10. Secondary Outcome: Mood State
Time Frame: baseline, 6, 12, 18, and 30 months
Reporting Status: Not Posted

11. Secondary Outcome: Physical Activity, Energy Expenditure
Description: change from baseline in energy expenditure at 12 months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: kcal/wk
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 85 | 94
kcal/wk | 814.8 (141.0) | 554.6 (134.9)

12. Secondary Outcome: Physical Activity, Energy Expenditure
Description: change from baseline in energy expenditure at 18 months
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kcal/wk
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 77 | 81
kcal/wk | 856.3 (177.6) | 356.0 (189.9)

13. Secondary Outcome: Change From Baseline in Energy Intake at 12months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 85 | 94
kcal/day | -544.1 (80.7) | -538.2 (78.2)

14. Secondary Outcome: Change From Baseline in Energy Intake at 18 Months
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Number analyzed (Participants) | 77 | 81
kcal/day | -326.3 (128.7) | -490.1 (134.0)

15. Secondary Outcome: Waist-to-hip Ratio at 6 Months
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Women SBT and MTT | Men SBT and MTT
Number analyzed (Participants) | 113 | 100
ratio | .84 (.01) | .96 (.01)

16. Secondary Outcome: Waist-to-hip Ratio at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Women SBT and MTT | Men SBT and MTT
Number analyzed (Participants) | 113 | 100
ratio | .83 (.01) | .95 (.01)

17. Secondary Outcome: Waist-to-hip Ratio at 18 Months
Time Frame: 18 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Women SBT and MTT | Men SBT and MTT
Number analyzed (Participants) | 113 | 100
ratio | .83 (.01) | .96 (.01)

18. Secondary Outcome: Waist-to-hip Ratio at 30 Months
Time Frame: 30 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Women SBT and MTT | Men SBT and MTT
Number analyzed (Participants) | 113 | 100
ratio | .85 (.01) | .97 (.01)

ADVERSE EVENTS:
Arm/Group | Standard Behavioral Treatment (SBT) | Maintenance-Tailored Treatment (MTT)
Serious Adverse Events (participants affected / at risk) | 0/106 | 1/107
Other Adverse Events (participants affected / at risk) | 29/106 | 26/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Behavioral Treatment (SBT) (N=106) | Maintenance-Tailored Treatment (MTT) (N=107)
heart attack death (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Behavioral Treatment (SBT) (N=106) | Maintenance-Tailored Treatment (MTT) (N=107)
cardiac events (Cardiac disorders) | 4 (4) | 3 (3)
Skin event (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
musculoskeletal events (Musculoskeletal and connective tissue disorders) | 12 (12) | 13 (13)
surgical events (Surgical and medical procedures) | 3 (3) | 3 (3)
ear event (Ear and labyrinth disorders) | 0 (0) | 1 (1)
gastrointestinal events (Gastrointestinal disorders) | 1 (1) | 2 (2)
endocrine events (Endocrine disorders) | 1 (1) | 0 (0)
pregnancies (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
reproductive events (Reproductive system and breast disorders) | 1 (1) | 1 (1)
infection (Infections and infestations) | 1 (1) | 0 (0)
renal event (Renal and urinary disorders) | 1 (1) | 1 (1)
eye events (Eye disorders) | 1 (1) | 1 (1)
skin event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No